CLINICAL TRIAL: NCT06123351
Title: Forward Head Posture Correction Impact on Temporomandibular Dysfunction: A Randomized Controlled Trial
Brief Title: Forward Head Posture Correction Impact on Temporomandibular Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shima Abdollah Mohammad Zadeh (Other)
Responsible Party: Sponsor-Investigator, Shima Abdollah Mohammad Zadeh, Principal Investigator, University of Sharjah
Organization: University of Sharjah (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FHP-TMD
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Temporomandibular Disorder; Forward Head Posture
Keywords: Traction; Exercise; Pain; Temporomandibular dysfunction
MeSH Terms: conditions — Temporomandibular Joint Disorders; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: Permuted block randomization to ensure an equal number of allocations in each of the three groups (traditional, Denneroll cervical traction orthodontic and dental treatment). Each random block was stored in opaque sealed envelopes consecutively numbered with a third researcher. Once each participant officially joins the study the researcher will open the subsequent envelop.
Who Masked: Participant
Masking Description: Single blinded study where the participants will be blinded to the study different groups and the study hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Denneroll protocol (Experimental): orthotic will be placed under participants' neck. Treatment session time begin with 3 minutes then increase of 2-3 minutes until they reach 15 to 20 minutes in each session.
  Interventions: Device: Denneroll cervical traction orthodontic
- Traditional protocol (Active Comparator): consists of one strengthening exercise for 10 repetitions in 3 sets each, and two stretching exercises with a hold for 20-30 seconds.
  Interventions: Other: stretching and strengthening exercises
- Dental management (Active Comparator): formed soft occlusal splint will be individually designed for the upper arch of each participant.
  Interventions: Device: Vacuum-formed soft occlusal splint

INTERVENTIONS:
Device: Denneroll cervical traction orthodontic — traction for 3 to 15 minutes once daily
  Arms: Denneroll protocol
Other: stretching and strengthening exercises — strengthening exercises with 10 repetitions twice per day 3 times per week stretching exercises with hold for 20 to 30 seconds 3 repetitions daily
  Arms: Traditional protocol
Device: Vacuum-formed soft occlusal splint — 2 mm thick elastic rubber sheets
  Arms: Dental management

SUMMARY:
The goal of this clinical trial is to test the effect of nerd neck correction on damaged jaw in people who suffers from jaw problems and nerd neck. The main question it aims to answer:

* whether there are different effects of traditional nerd neck correction exercises, device correction method and dental splints on jaw features of pain and function.

Participants will:

* participants will be given the consent to sign first.
* participants will be assessed to check jaw pain and function.
* participants will be divided randomly into 3 groups.
* Each group will be given the treatment sessions for 6 weeks.
* participants will come back after 6 weeks for one last assessment.

Researchers will compare traditional, new and dental treatment groups to see if there is improvement in jaw characteristics.

DETAILED DESCRIPTION:
The relationship between the two conditions of forward head posture (FHP) and temporomandibular joint dysfunction (TMD) have been previously stated with comparing the craniocervical angle (CVA) of TMD patients to the healthy individuals, still a clear relationship couldn't be drawn due to different study limitations such as the lack of subdivision in the TMD patients based on their diagnostic subcategories in addition to, patients posture might have been altered while the photo was captured. Ever since, multiple researchers deliberately investigated the two conditions association and inferred the following: 1. FHP can be a risk factor resulting in TMD where any alteration in the head position produces more tension on the masticatory muscles by changing the mandible position 2. TMD origins from muscular component is more significant than articular component yet the correlation between head posture and TMD is still not clear enough, however, if FHP and myogenic TMD were linked preventive measures can be taken. recently, multiple studies established a relation between the occurrence of FHP in TMD patients which supported the hypothesized relation between them.

Till present, no study has investigated the FHP Denneroll cervical traction orthodontic (DCTO) correction impact alone on TMD and this is where the purpose of this study arises from.

ELIGIBILITY:
Inclusion Criteria:

* The participant experiencing one or more of TMD signs or symptoms and has been diagnosed with TMD beside having forward head posture with craniocervical (CVA) angle < 50.
* The study will be limited to the patients in the dental clinic of the university of Sharjah.
* Participants experiencing mild to moderate myogenic TMD with symptoms of orofacial pain and limited range of jaw opening.

Exclusion Criteria:

* Previous head, neck or TMJ traumas.
* History of temporomandibular joint surgery.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Anamnestic questionnaire by Fonseca | Baseline (pre-treatment) and week 7 (post-treatment)
  To evaluate TMD by 10 questions with their corresponding scores from 0 to 1
Craniocervical angle - CVA | Baseline (pre-treatment) and week 7 (post-treatment)
  photographic method to evaluate the angle where an angle less than 50 degrees will be considered as forward head posture

SECONDARY OUTCOMES:
Boley Gauge | Baseline (pre-treatment) and week 7 (post-treatment)
  Electronic Digital Caliper to assess mouth opening (active/passive)
Numerical Rating Scale (NRS) | Baseline (pre-treatment) and week 7 (post-treatment)
  0-10 scale (zero represents no pain and 10 is the worst pain ever) to record orofacial pain
Mandibular Opening | Baseline (pre-treatment) and week 7 (post-treatment)
  Tape to measure the distance between the incisal edges of upper and lower teeth

CONTACTS AND LOCATIONS:
Overall Officials: Shima Mohammad zadeh, Study Director — University of Sharjah; Tamer Shousha, Principal Investigator — University of Sharjah
Locations (1):
- University of Sharjah, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Lee WY, Okeson JP, Lindroth J. The relationship between forward head posture and temporomandibular disorders. J Orofac Pain. 1995 Spring;9(2):161-7. PMID 7488986
- [Background] Salkar RG, Radke UM, Deshmukh SP, Radke PM. Relationship between temporomandibular joint disorders and body posture. Int J Dent Health Sci. 2015;2(6):1523-30.
- [Background] Saddu SC, Dyasanoor S, Valappila NJ, Ravi BV. The Evaluation of Head and Craniocervical Posture among Patients with and without Temporomandibular Joint Disorders- A Comparative Study. J Clin Diagn Res. 2015 Aug;9(8):ZC55-8. doi: 10.7860/JCDR/2015/12830.6343. Epub 2015 Aug 1. PMID 26436048
- [Background] El-Hamalawy FA. Forward head correction exercises for management of myogenic tempromandibular joint dysfunction. 2011;7(8)
- [Background] Tang Y, Xu LL, Fan S. [Control study of forward head posture between patients with temporomandibular disorders and healthy people]. Shanghai Kou Qiang Yi Xue. 2021 Apr;30(2):173-176. Chinese. PMID 34109357
- [Background] Xiao CQ, Wan YD, Li YQ, Yan ZB, Cheng QY, Fan PD, Huang Y, Wang XY, Xiong X. Do Temporomandibular Disorder Patients with Joint Pain Exhibit Forward Head Posture? A Cephalometric Study. Pain Res Manag. 2023 Feb 2;2023:7363412. doi: 10.1155/2023/7363412. eCollection 2023. PMID 36776487
- [Background] Minervini G, Franco R, Marrapodi MM, Crimi S, Badnjevic A, Cervino G, Bianchi A, Cicciu M. Correlation between Temporomandibular Disorders (TMD) and Posture Evaluated trough the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD): A Systematic Review with Meta-Analysis. J Clin Med. 2023 Apr 2;12(7):2652. doi: 10.3390/jcm12072652. PMID 37048735